CLINICAL TRIAL: NCT05238805
Title: Double Pet Project : A Comparison Between 11C-Acetate and 11C-acetoacetate Heart and
Brief Title: Double Pet Project : A Comparison Between 11C-Acetate and 11C-acetoacetate Heart and Kidney Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-4540
Record Dates: First submitted 2022-01-04; First posted 2022-02-14 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Ketoses, Metabolic
Keywords: ketones; heart metabolism; kidney metabolism
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Participants will have to perform 2 scans one after the other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational heart and kidney metabolism (Other): Participants will have a PET scan with 11C-Acetate followed by a TEP Scan with 11C-Acetoacetate all in the same day.
  Interventions: Radiation: Observational heart and kidney on siemens TEP scan

INTERVENTIONS:
Radiation: Observational heart and kidney on siemens TEP scan — Same as arm description

SUMMARY:
The objective of this study is to make a comparison between 11C-acetate and 11C-Acetoacetate heart and kidney metabolism

DETAILED DESCRIPTION:
Healthy people will have two positron emission tomography scan to perform. One, with a 11C-Acetate Tracer and the other with 11C-Acetoacetate. The results will allow to determine if both tracers are used in a similar way but the organs and see if the investigators can use the already validated analyse method for acetate to make acetoacetate analysis

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55
* BMI between 18,5 and 28
* Healthy
* Normal value for blood pressure

Exclusion Criteria:

* Taking drugs that could influence metabolism
* Diabetes or prediabetes
* Pregnancy or lactation
* Participation in a intensive sport program
* Being on a ketogenic diet
* Any clinical abnomally in prescreen blood sample

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
Mean in left ventricule myocradial blood flow | 30 minutes
  Heart acetate metabolism measured by TEP scan
Mean in left ventricule myocardial blood flow | 30 minutes
  Heart acetoacetate metabolism measured by TEP scan
Mean in Kidney acetate uptake | 30 minutes
  Kidney acetate uptake measured by TEP scan
Mean in Kidney acetoacetate uptake | 30 minutes
  Kidney acetoacetate uptake measured by TEP scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada